CLINICAL TRIAL: NCT03985254
Title: Does Adding Power Exercises to Muscle Force Training Result in Superior Benefits for Patellofemoral Pain People? Randomized and Controlled Clinical Trial
Brief Title: Do Power Exercises Result in Superior Benefits for People With Patellofemoral Pain?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Gabriela Souza de Vasconcelos, Post graduate, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LaiotUFSCAR
Record Dates: First submitted 2019-06-10; First posted 2019-06-13 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strength Training Group (STG) (Active Comparator): The strength training program will consist of applying resistance and progressive exercises for strength gain and will be based on the training principles recommended by the American College of Sport Medicine. The exercises were chosen based on a pilot study that successfully applied the protocol to 10 participants with FPD (data to be published) and other strength training studies (MASCALL et al, 2003; DISTEFANO et al, 2009; REIMAN et al, 2012; BALDON et al, 2014; SILVA et al, 2015).
  Initially, the goal will be the development of neuromotor control and resistance (load <50% of the one repetition maximum test [1RM]), and in subsequent weeks the goal will be the development of muscle strength (load> 70% 1RM). In addition, the protocol will initially focus on strengthening the hip and trunk muscles and after four weeks of training, exercises for the knee muscles will be included.
  Interventions: Other: Strength Training Group (STG)
- Strength and Power Training Group (SPTG) (Experimental): Participants who are allocated to this group will perform the same exercise program performed by the STG, but with the addition of exercises that emphasize power gain. As in the other group, initially, the objective will be the development of neuromotor control and resistance (load <50% of the one repetition maximum test [1RM]). However, in subsequent weeks the goal will be to develop strength (load> 70% 1RM) and muscle power (load between 40-60% 1RM).
  Interventions: Other: Strength and Power Training Group (SPTG)

INTERVENTIONS:
Other: Strength Training Group (STG) — The strength training program will consist of applying resistance and progressive exercises for strength gain and will be based on the training principles recommended by the American College of Sport Medicine. The exercises were chosen based on a pilot study that successfully applied the protocol to 10 participants with FPD (data to be published) and other strength training studies (MASCALL et al, 2003; DISTEFANO et al, 2009; REIMAN et al, 2012; BALDON et al, 2014; SILVA et al, 2015).
  Initially, the goal will be the development of neuromotor control and resistance (load <50% of the one repetition maximum test [1RM]), and in subsequent weeks the goal will be the development of muscle strength (load> 70% 1RM). In addition, the protocol will initially focus on strengthening the hip and trunk muscles and after four weeks of training, exercises for the knee muscles will be included.
  Arms: Strength Training Group (STG)
Other: Strength and Power Training Group (SPTG) — Participants who are allocated to this group will perform the same exercise program performed by the STG, but with the addition of exercises that emphasize power gain. As in the other group, initially, the objective will be the development of neuromotor control and resistance (load <50% of the one repetition maximum test [1RM]). However, in subsequent weeks the goal will be to develop strength (load> 70% 1RM) and muscle power (load between 40-60% 1RM).
  Arms: Strength and Power Training Group (SPTG)

SUMMARY:
Patellofemoral pain (PFP) is one of the most common forms of knee pain and has a negative impact on the level of physical activity and quality of life of patients. Although strengthening of the hip and knee muscles has good clinical effects in the treatment of PFP, most exercise protocols do not follow the American College of Sports Medicine (ACSM) guidelines and are not clearly described, making it difficult to apply them in practice clinical and research. In addition, recent studies have shown that these patients also have a power deficit of these muscles. However, it is not known whether the addition of power exercises to a muscle strengthening program would result in superior benefits, especially in relation to pain and physical function. Therefore, the objective of this study is to verify if the improvement in pain intensity, physical function, kinesiophobia, self perception of improvement, quality of life and muscle function variables after a training program of strength and muscular power is superior to that observed in an isolated muscle strength training. This study will be randomized and controlled, developed with individuals with DPF, allocated in one of two groups: Strength Training Group (STG) and Strength and Power Training Group (SPTG). The primary outcomes will be intensity of pain and physical function, while the secondary outcomes will be kinesiophobia; self perception of improvement; quality of life; the peak of isometric abductor and hip extensor torque, and knee extensor; and the rate of development of torque of the abductors and extensors of hip, and extensors of knee at 30% and 90% of maximum isometric torque. Participants in both groups will be evaluated before the intervention (pre), after the end of the intervention (post) and three, six and twelve months after the intervention. Data analysis will follow the intention-to-treat principle. To compare the groups at different times (pre, post and after three, six and twelve months of the intervention) will be used two-way analysis of variance (GROUP X MOMENT) with mixed model, with Bonferroni post hoc to identify specific differences. The significance level will be 0.05.

ELIGIBILITY:
Inclusion Criteria:

* men and women with bilateral or unilateral patellofemoral pain

Exclusion Criteria:

* history of knee surgery
* history of hip or lumbar spine injury or pain
* patellar instability
* pain on palpation of the patellar tendon, iliotibial band, Hoffa fat, goose paw tendons or knee joint line
* signs or symptoms of meniscal or knee ligament injuries
* presence of Osgood-Schlatter syndrome or Sinding-Larsen-Johansson syndrome
* any vestibular, neurological or musculoskeletal alterations that interfere or contraindicate the procedures of this study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline pain Intensity at 12 weeks | Pre (baseline) treatment, post treatment (12 weeks) and after 3,6 and 12 month (follow-up)
  Pain intensity will be assessed using a 100-mm Visual Analog Scale (VAS), with 0 indicating no pain and 10 indicating extremely intense pain. Participants will indicate their usual pain and their worst pain during the last week (CROSSLEY et al, 2004). The VAS scores will be computed by measuring the length of the line, in millimeters, from the left end (without pain) until the mark made by the participant.
Change from baseline physical function at 12 weeks | Pre (baseline) treatment, post treatment (12 weeks) and after 3,6 and 12 month (follow-up)
  The Anterior Knee Pain Scale, a translated and validated Portuguese version (DA CUNHA et al, 2013), will be used to evaluate subjective symptoms, such as anterior knee pain and functional limitations related to PFP. The items assessed in the questionnaire are patellar subluxation, lameness, pain, walking, climbing stairs and remaining seated for prolonged time with knees flexed. It has scores of 0 to 100 points, where 100 means no pain and / or functional limitations and 0 means constant pain and several functional limitations (KUJALA et al, 1993). The Anterior Knee Pain Scale is a reliable and valid instrument to evaluate the function in individuals with PFP (CROSSLEY et al, 2004). The final score will be used for statistical analysis.

SECONDARY OUTCOMES:
Kinesiophobia | Pre (baseline) treatment and post treatment (12 weeks)
  The kinesiophobia will be assessed using the translated and validated version of the Tampa Scale for Kinesiophobia questionnaire (SIQUEIRA et al, 2007), which is composed of 17 items that evaluate fear of movement, injury or recurrence of injury (MILLER, 1991). This questionnaire is a four-point Likert scale, in which the sum of responses can vary from 17 to 68, and scores greater than 37 indicate the presence of kinesiophobia.
Self-perception of improvement | Pre (baseline) treatment and post treatment (12 weeks)
  The global rating of change (GRC) scale is a 15-point, single-item scale that measures the patient's im¬pression of improvement in health status following treatment (JAESCHKE et al, 1989). The scale is scored from -7 (a very great deal worse) to +7 (a very great deal better), with 0 (zero) indicating that there was no change. Changes of 4 points or more in this scale were previously considered to be clinically important in patients with knee pain.
Change Quality of Life | Pre (baseline) treatment and post treatment (12 weeks)
  Participants' quality of life will be assessed through the Knee Injury and Osteoarthritis Outcome Score (KOOS). This questionnaire is composed of 42 items, divided into 5 sub-scales, which assess: pain, symptoms, function in sports and recreational activities, function in daily life activities and quality of life in adults with knee injuries (ligaments, meniscal) including post-traumatic osteoarthrosis. In the present study, only the sub-scale of quality of life will be applied to participants. This sub-scale is composed of four questions and each one will be scored from 0 to 4, 0 representing extreme knee problems and 4 that there are no problems in the knee. The sum of these questions will be used for further analysis.
Maximal Isometric Torque and Rate of Force Development (RFD) | Pre (baseline) treatment and post treatment (12 weeks)
  The maximal isometric torque of the hip abductors and extensors, and knee extensors, as the rate of force development, will be assessed using an isokinetic dynamometer (Biodex MultiJoint System 3, Biodex Medical Systems Inc., New York, USA), with a sampling frequency of 100 Hz.
  To calculate the RFD of the hip abductors and extensors and knee extensors, the data of the repetitions in which the participants reached the highest isometric torque will also be used (NUNES et al, 2018). The normalized torque data will be exported and processed in Matlab software.
  The evaluation of the RFD will be performed by calculating the slope of the torque/time curve. The slope will be obtained by dividing the normalized torque variation (Nm/kg × 100, represented as %) by the time variation (ms) from the start of the contraction until 30% and 90% of the maximal isometric torque (BELLEW, 2002; CHANG et al, 2005).

CONTACTS AND LOCATIONS:
Locations (1):
- Gabriela Souza de Vasconcelos, São Carlos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vasconcelos GS, Nunes GS, Munhoz RF, da Silva MECB, Pisani GK, Luz BC, Serrao FV. Is strength and power training targeting hip and knee muscles superior to strength training in individuals with patellofemoral pain? Proof of concept study. Sci Rep. 2024 Nov 10;14(1):27450. doi: 10.1038/s41598-024-78074-2. PMID 39523423
- [Derived] de Vasconcelos GS, Nunes GS, Barton CJ, Munhoz RF, da Silva MECB, Pisani GK, Luz BC, Serrao FV. Adding muscle power exercises to a strength training program for people with patellofemoral pain: protocol of a randomized controlled trial. Trials. 2021 Nov 6;22(1):777. doi: 10.1186/s13063-021-05748-x. PMID 34742328